CLINICAL TRIAL: NCT06780891
Title: Telephysical Therapy as a Secondary Stroke Prevention Tool
Brief Title: Effectiveness of Telephysical Therapy as a Secondary Stroke Prevention Tool in Patients With Minor Stroke.
Acronym: TPT-Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Collaborators: Hospital Universitario Virgen Macarena (Other)
Responsible Party: Principal Investigator, Ignacio Pastor Ruiz, Principal Investigator, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0616-N-22
Record Dates: First submitted 2025-01-10; First posted 2025-01-17 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Physical Therapy Modality; Secondary Prevention; Physical Therapy Evaluation; Therapeutic Exercise; Randomized Controlled Trial; Cerebrovascular Accident (Stroke)
Keywords: Ischemic Attack, Transient; Brain Ischemia; Telephysical Therapy; Exercise Therapy; Neurological Disorders; Wearable Electronic Devices; Quality of life
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Brain Ischemia; Nervous System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telephysical therapy group with educational session (Experimental): The intervention includes 12 weeks of therapeutic exercise delivered via tele-assistance. Participants will engage in aerobic and anaerobic activities focusing on cardiovascular fitness, muscle strength, and balance. A recorded educational session will provide uniform information on the protocol, including schedules and intervention details. Patients will complete prescribed exercises under virtual supervision and submit progress reports for monitoring adherence.
  Interventions: Behavioral: Telephysical therapy; Behavioral: Educational session
- Educational session with encouraged lifestyle modifications (Active Comparator): The control group will be encouraged to return to their regular daily activities and engage in exercise. Evaluations will be scheduled and communicated to participants. The control group will not receive direct intervention.
  Interventions: Behavioral: Educational session

INTERVENTIONS:
Behavioral: Telephysical therapy — The experimental group is undergoing a tele-assisted therapeutic exercise program (T-TPT/T-FIS), which involves physical exercises aimed at improving cardiovascular fitness, muscle strength, and balance, among others. Participants will complete exercises under virtual supervision and submit progress reports.
  Arms: Telephysical therapy group with educational session
Behavioral: Educational session — The educational session will focus on raising awareness about stroke risk factors, such as hypertension, diabetes, and smoking, while promoting healthy lifestyle changes. The goal is to empower them with the knowledge to reduce stroke risk and improve overall well-being.

SUMMARY:
This study investigates the effectiveness of telephysiotherapy as a rehabilitation and secondary prevention tool in patients with minor stroke, TIA, or LACI, comparing an experimental group receiving tele-assisted aerobic and anaerobic exercises to a control group.

DETAILED DESCRIPTION:
Stroke is an acute disorder of cerebral blood flow that can cause transient or permanent alterations in the functionality of the brain, often resulting from ischemia or hemorrhage. Depending on the affected region and its severity, strokes range in impact, with minor strokes characterized by mild symptoms. Despite the potential for rapid symptom improvement in transient ischemic attacks (TIAs), both minor strokes and TIAs significantly impact long-term quality of life.

The implementation of physical rehabilitation, particularly through structured exercise, is critical for mitigating motor deficits, reducing fatigue, and improving functional capabilities post-stroke. Tele-physical therapy (TPT)/Therapeutic Tele-Assisted Exercise (T-TEx/T-FIS) has emerged as a promising approach for delivering rehabilitation remotely, offering convenience and ensuring continuity of care while addressing limitations posed by traditional in-person therapy. Recent systematic reviews suggest that TPT/T-TEx/T-FIS demonstrates comparable outcomes to conventional physiotherapy, highlighting its potential for wider adoption.

The hypothesis is that a 12-week tele-physiotherapy program can significantly improve cardiovascular health, reduce obesity, and enhance quality of life in patients with minor stroke, TIAs, or lacunar infarcts, compared to standard lifestyle recommendations alone. The primary objective is to evaluate the efficacy of tele-physiotherapy in addressing modifiable risk factors for secondary stroke prevention. Secondary goals include analyzing improvements in cardiorespiratory fitness, muscle strength, sleep quality, and fatigue, while promoting healthy lifestyle habits and tracking adherence to therapeutic exercise.

A single-blind, randomized controlled trial is proposed, wherein patients are divided equally into a control group and an experimental group receiving TPT. Participants will undergo assessments at baseline, 4 weeks, and 12 weeks, with a follow-up at 24 weeks to evaluate sustained benefits.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Subjects with a diagnosis of minor stroke, TIA, or LACI immediately after hospital discharge.
* Age: Between 35 and 85 years.
* Technology access: Ownership of a smartphone with Android operating system and internet access.
* Language skills: Ability to read, write, and understand instructions in Spanish, or the presence of a caregiver who can perform these tasks on behalf of the patient.
* Motor impairment: Minimal motor sequelae, defined by:
* "Timed Up and Go" (TUG) test: In less than 13.5 seconds.
* Score of 3-5 points on the Functional Ambulatory Category (FAC).
* Walking capacity: Ability to walk independently for 500 meters without technical or physical assistance.
* Spasticity: Minimal or absent spasticity (score of 0-1 on Ashworth Scale

Exclusion Criteria:

* Oxygen dependency: Dependency on auxiliary oxygen.
* Uncontrolled or unstable conditions: Including angina pectoris, hypertension (defined as resting systolic blood pressure >180 mm Hg and diastolic >110 mm Hg), arrhythmias (atrial/ventricular), sinus tachycardia (heart rate >120/min), and diabetes mellitus.
* Orthostatic hypotension: Drop in blood pressure >20 mm Hg with associated symptoms.
* Significant aortic stenosis: Defined as a diameter <1 cm², or aortic dissection.
* Uncompensated cardiac failure: Including third-degree atrioventricular block without a pacemaker, active myocarditis/pericarditis, and atrial fibrillation.
* Recent embolism: Pulmonary or systemic embolism, or acute thrombophlebitis.
* Systemic illness or fever: Presence of acute systemic disease or fever.
* Musculoskeletal conditions: That prevent participation in the therapeutic exercise program.
* Other metabolic conditions: Such as acute thyroiditis, hypo/hyperkalemia, and hypovolemia (until treated).
* Severe psychological disorders: Diagnosed severe psychological conditions.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Quality of life (SF-36) | Initial baseline assessment (week 1), assessment post-intervention (week 12) and assessment post-intervention 2 (week 24).
  Assessed using the SF-36 questionnaire, which evaluates physical and mental health domains. The scale consists of 36 questions, assesing physical function (10 items), physical role (4 items), bodily pain (2 items), general health status (5 items), vitality (4 items), social function (2 items), emotional role (3 items), mental health (5 items), and health transition (1 item). A higher score indicates better health status.
Gait characteristics (GAITRite system and 6MWT) | Initial baseline assessment (week 1), assessment post-intervention (week 12) and assessment post-intervention 2 (week 24).
  Assessed using the GAITRite system and the 6-minute walk test (6MWT). The GAITRite system will measure weight distribution, support surface, time in double support and single support, step time, step symmetry and length, and gait normality. Measurements will be taken while wearing shoes, both before and after performing the 6MWT. The 6-minute walk test (6MWT) is a validated test and is considered highly reliable for measuring gait in stroke patients. Additionally, its execution has been validated in environments with limited space (15 and 30 meters), making it easier to use. It will also allow us to assess the response to exertion, as well as the gait adjustments associated with fatigue.
Fall risk and functional mobility (TUG) | Initial baseline assessment (week 1), assessment post-intervention (week 12) and assessment post-intervention 2 (week 24).
  Asesssed using the Timed Up and Go (TUG) Test. It is a valid, reliable, and easy-to-administer fall risk test used to measure advanced functional mobility after a stroke. To perform this test, the patient must rise from a chair, walk three meters, and return to sit as quickly as possible.
Balance (BBS) | Initial baseline assessment (week 1), assessment post-intervention (week 12) and assessment post-intervention 2 (week 24).
  Assessed using the Berg Balance Scale (BBS), which is designed to evaluate balance and predict gait and fall risk. This scale complements the Timed Up and Go (TUG) test. It includes 14 tasks, with the patient's movement quality rated on a scale from 0 to 4. The maximum achievable score is 56/56.
Walking and assistance (FAC) | Initial baseline assessment (week 1), assessment post-intervention (week 12) and assessment post-intervention 2 (week 24).
  Assesed using the level of walking and assistance using the Functional Ambulation Classification (FAC) Scale . This scale evaluates the patient's walking capacity and the degree of support required, categorizing walking ability into six distinct levels.
Fatigue associated with stroke (FSS) | Initial baseline assessment (week 1), assessment post-intervention (week 12) and assessment post-intervention 2 (week 24).
  Assessed the level of fatigue related to the stroke using the Fatigue Severity Scale. It is a 9-item scale that captures the patient's subjective assessment of their fatigue and its impact on their life, with scores ranging from 1 to 7. The possible values range from 9 to 63, with a lower score indicating a better outcome.
Handgrip strength (Digital Dynamometer) | Initial baseline assessment (week 1), assessment post-intervention (week 12) and assessment post-intervention 2 (week 24).
  Measured to assess muscular strength and serves as a predictor of cardiovascular events, chronic diseases, and overall health. Studies highlight its predictive value. A digital dynamometer from the brand Vicfund will be used for its measurement.

SECONDARY OUTCOMES:
Body mass index (BMI) | Initial baseline assessment (week 1), assessment post-intervention (week 12) and assessment post-intervention 2 (week 24).
  Weight and heigh will be combined to report Body Mass Index (BMI). While BMI is a useful health indicator for any patient, its influence on stroke has also been documented. Data will be collected using a tape measure and a scale. It will be recorded in kg/m^2.
Sagittal abdominal diameter (SAD) | Initial baseline assessment (week 1), assessment post-intervention (week 12) and assessment post-intervention 2 (week 24).
  Abdominal fat accumulation is a key component of the cardiometabolic syndrome, which is associated with stroke, heart attack, cardiovascular diseases, metabolic complications, and overall mortality. It has been shown that this risk increases when the diameter exceeds 25 cm. Data will be collected using a tape measure. It will be recorded in cm.
VO2 peak | Initial baseline assessment (week 1), assessment post-intervention (week 12) and assessment post-intervention 2 (week 24).
  VO2 peak will allow us to assess cardiorespiratory health. It will be measured using a smartwatch while the patient is lying down, 5 minutes after exercise. It will be recorded in ml O2/kg/min.
Blood pressure | Initial baseline assessment (week 1), assessment post-intervention (week 12) and assessment post-intervention 2 (week 24).
  Blood pressure will be measured in a seated position before exertion, after exercise, and 5 minutes post-rest, using a smartwatch. The value will be recorded in mmHg.
Biochemical levels | Initial baseline assessment (week 1), assessment post-intervention (week 12) and assessment post-intervention 2 (week 24).
  These are considered the main modifiable risk factors for stroke recurrence. Blood lipid and glucose levels will be collected through biochemical analysis provided by the hospital's blood collection service. The sample will be taken on the same day as the evaluation, with analysis and result collection afterward. Patients should fast for a minimum of 8 to 12 hours before the extraction, as is also required for blood pressure measurement.
  * Glucose: Measured in mg/dl, and consideration will be given to whether the patient has diabetes mellitus. Additionally, glycated hemoglobin will be recorded.
  * Lipids: The following lipid parameters will be measured: LDL (low-density lipoprotein), HDL (high-density lipoprotein), total cholesterol, and triglycerides.
Adherence to therapy | Daily throughout the duration of the study (from baseline (week 1) to post-intervention 2 (week 24)).
  Assessed through an online form. The patient will complete a daily Google form where they will record the values obtained from the smartwatch, alcohol, and tobacco consumption, as well as their subjective feelings of effort and rest. Adherence will be measured by the number of forms submitted throughout the study and the data provided in them.
Perceived exertion | Initial baseline assessment (week 1), assessment post-intervention (week 12) and assessment post-intervention 2 (week 24).
  To dose physical activity, understanding the sensation of exertion will allow us to program the workload more selectively for each patient. The Borg scale has proven useful for this purpose and is also easy for the patient to record. To use it, the patient simply needs to rate the level of fatigue associated with the exertion on a scale from 0 to 10.
Harmful habits and sleep | Daily throughout the duration of the study (from baseline (week 1) to post-intervention 2 (week 24)).
  Tobacco and alcohol consumption are recognized as risk factors for suffering from strokes. Therefore, it will be important to record this information to evaluate the evolution of the patient's habits and the impact of their consumption on other parameters. For measurement, the patient will manually record their consumption daily in a form, indicating "cigarettes consumed" and "glasses of alcoholic beverages."
  The subjective quality of sleep in post-stroke patients is related to depression and affects physical functionality. To measure this, the patient will rate the quality of their rest on a scale from 0 to 10 in the form daily and will also record the number of hours of sleep monitored by the smartwatch.

CONTACTS AND LOCATIONS:
Overall Officials: David Manuel Lucena Antón, Doctor of PT, Study Director — University of Cadiz
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Sevilla, Spain

IPD SHARING:
Plan to Share IPD: No